CLINICAL TRIAL: NCT00171080
Title: A 2 x 5-week Multicenter, Cross-over Study to Compare the Reduction of Predialysis Systolic Blood Pressure With Valsartan 80 mg Compared to Irbesartan 150 mg in Patients With Mild to Moderate Hypertension on Long-term Hemodialysis
Brief Title: VALID: Study to Compare the Reduction of Predialysis Systolic Blood Pressure With Valsartan Compared to Irbesartan in Patients With Mild to Moderate Hypertension on Long-term Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CVAL489ADE19
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Hypertension
Keywords: Hypertension; Valsartan; Dialysis; Renal Disease
MeSH Terms: conditions — Hypertension; Kidney Diseases | interventions — Valsartan; Irbesartan

INTERVENTIONS:
Drug: valsartan
Drug: irbesartan

SUMMARY:
The purpose of the study is to compare the efficacy, safety and tolerability of valsartan 80 mg (with a starting dose of 40 mg) to irbesartan 150 mg (with a starting dose of 75 mg) in patients on long-term haemodialysis with mild to moderate increased mean supine systolic blood pressure (MSSBP).

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild and moderate hypertension defined by a MSSBP ≥ 140 mmHG and < 180 mmHG at Visits 1 and 2 for treated and untreated patients
* Chronic hemodialysis for at least 6 months prior to Visit 1 as substitution therapy.
* If treated with epoetin: patients with a stable hematocrit ≤ 40% (± 5%).

Exclusion Criteria:

* Inability to discontinue angiotensin II receptor blockers (ARBs) safely for a period of 1 week, as required by the protocol.
* Treatment with more than 3 different compounds for the treatment of hypertension at Visit 1.
* Atrial fibrillation

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2004-04; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in systolic blood pressure after 4 weeks

SECONDARY OUTCOMES:
Change from baseline in diastolic blood pressure after 4 weeks
Systolic blood pressure less than 100 mmHg with or without symptoms of low blood pressure
Adverse events and clinical laboratory abnormal results
Change from baseline in average 24-hour ambulatory blood pressure after 4 weeks
Change from baseline in daytime and nighttime ambulatory blood pressures after 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Investigative Centers, Germany
- Novartis Pharmaceuticals, Basel, Switzerland

REFERENCES:
- [Result] Leidig M, Bambauer R, Kirchertz EJ, Szaba T, Handrock R, Leinung D, Baier M, Schmieder RE. Efficacy, safety and tolerability of valsartan 80 mg compared to irbesartan 150 mg in hypertensive patients on long-term hemodialysis (VALID study). Clin Nephrol. 2008 Jun;69(6):425-32. doi: 10.5414/cnp69425. PMID 18538118